CLINICAL TRIAL: NCT01277861
Title: Airway Responses During Desflurane Anesthesia Via a Laryngeal Mask Airway: Effects of Fentanyl Pretreatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Girish P Joshi, MD, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 092010-013
Record Dates: First submitted 2010-11-03; First posted 2011-01-17 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Administration Site Reaction
Keywords: Desflurane, Fentanyl, Airway responses
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FENTANYL (Active Comparator): FENTANYL
  Interventions: Drug: Fentanyl
- SALINE (Placebo Comparator): SALINE
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — FENTANYL PRETREATMENT DURING INDUCTION OF ANESTHESIA

SUMMARY:
The investigators plan to test the hypothesis that pretreatment with fentanyl prior to induction of anesthesia would result in reduce the incidence of movements and airway responses to desflurane in patients breathing spontaneously through a laryngeal mask airway (LMA). The primary aim of this study is to assess the effect of fentanyl pretreatment on the incidence of movement during induction of anesthesia. Secondary aim of the study is to evaluate the effects of titration of fentanyl according to the respiratory rate on the incidence of intraoperative respiratory events such as coughing, breath holding and laryngospasm.

DETAILED DESCRIPTION:
After obtaining approval from the institutional review board and informed consent, 100 patients, 18-64 years of age, scheduled for elective superficial and peripheral surgery of less than 2 h duration would be enrolled in this prospective, randomized, double-blind, placebo-controlled study. Patients will be randomly assigned to one of two anesthetic techniques according to a computer-generated random numbers table. Patients will receive either fentanyl or saline prior to induction of anesthesia, while the rest of the anesthetic and analgesic technique will be standardized for all patients.

Exclusion criteria will include obesity (body mass index >30), pregnancy, history of gastroesophageal reflux, hiatal hernia, significant cardiovascular, pulmonary (e.g., reactive airway disease), hepatic, renal, neurologic, metabolic, and endocrine disease as well as history of alcohol and drug abuse as well as those requiring tracheal intubation.

After premedication with midazolam 2 mg, patients will be transferred to the operating room. On arrival in the operating room standard monitors and the BIS (BiSpectral Index)monitor will be applied. Patients will then be preoxygenated for 2-3 minutes with 100% oxygen, which will be followed by administration of either fentanyl 1 µg/kg (made up to 10 ml saline) or 10 ml saline (prepared by a person not involved in the study). Induction of anesthesia will be performed 2-3 minutes after administration of the study drug with propofol 2.0 - 2.5 mg/kg after lidocaine 2% 20-30 mg. After loss of eyelash reflex an appropriate size LMA will be placed. If the patients become apneic, manual ventilation will be performed with oxygen/nitrous oxide and desflurane, 3% dialed concentration initially and then titrated to maintain the BIS value of 50-60.

Anesthesia will be maintained with desflurane titrated to achieve a BIS value of 50-60, along with 50% nitrous oxide and oxygen. Once spontaneous breathing resumes, fentanyl 25-50 µg will be administered to achieve a respiratory rate of 10-15 breaths/minute. Additional propofol/fentanyl will be administered, if deemed necessary by the attending anesthesiologist. All patients will receive dexamethasone 4 mg, IV after induction of anesthesia and ondansetron 4 mg 20-30 minutes prior to the end of surgery. Desflurane will be discontinued after closure of the surgical wound.

A blinded observer will record patient demographics (age, weight, height) and history of smoking from preoperative evaluation. Data collected during the intraoperative period will include need for manual ventilation and duration of manual ventilation, duration of anesthesia, total doses of propofol and fentanyl, and time from discontinuation of desflurane until patient first follows verbal command as well as heart rate (HR), mean arterial blood pressure (MAP), end-tidal carbon dioxide, oxygen saturation, and end-tidal gas concentration will be recorded every 15 minutes.

Data collected in the postoperative period will include verbal rating score (0 to 10) will be used to assess pain, nausea, and vomiting in the recovery room every 15 minutes for one hour as well as the need for rescue medications will also be recorded.

Patients will also be contacted approximately 24 hours after surgery to evaluate their post operative course including occurrence of any adverse events. The patient will remain in the study for approximately 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years of age
* Subjects scheduled for elective superficial and peripheral surgery of less than 2 h duration (e.g., hernia surgery, breast surgery, upper or lower limb surgery, superficial abdominal/chest wall surgery [i.e., lipoma], minor gynecological procedures [i.e., hysteroscopy])

Exclusion Criteria:

* obesity (body mass index >30)
* pregnancy
* history of gastroesophageal reflux, hiatal hernia, significant cardiovascular, pulmonary (e.g., reactive airway disease), hepatic, renal, neurologic, metabolic, and endocrine disease
* history of alcohol and drug abuse
* requiring tracheal intubation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Girish P Joshi, MD, Principal Investigator — University of Texas Southwestern Medical Center, Dallas
Locations (1):
- Ut Southwestern Medical Center At Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited for the study in the preoperative period.
Pre-assignment Details: Participants were included based on inclusion/exclusion criteria. Participants were excluded if muscle relaxation was necessary for the surgery.
Period: Overall Study
Arm/Group | FENTANYL | SALINE
Started | 51 | 49
Completed | 49 | 47
Not Completed | 2 | 2
Not completed — Physician Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FENTANYL | SALINE | Total
Number analyzed (Participants) | 49 | 47 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 47 | 96
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 24 | 22 | 46
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Body mass index is calculated from height and weight of the patient.
  kg/m2 | 26.8 (4.3) | 26.8 (4.7) | 26.8 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Movement
Description: The data provided below include participants who moved (includes all grades of movement ie, mild, moderate and severe).
Time Frame: Induction of Anesthesia
Population: Per protocol
Measure: Number; unit: Participants, number
Groups:
- Fentanyl Pretreatment Group: Fentanyl 1 µg/kg (constituted to 10 ml with saline) prior to induction of anesthesia.
- Saline Pretreatment Group: Saline 10 ml prior to induction of anesthesia.
Arm/Group | Fentanyl Pretreatment Group | Saline Pretreatment Group
Number analyzed (Participants) | 49 | 47
Participants, number | 8 | 24

2. Secondary Outcome: Apnea
Description: Apnea defined as no breathing for at least 30 s.
Time Frame: Induction of Anesthesia
Population: Per protocol
Measure: Number; unit: Participants, number
Arm/Group | Fentanyl Pretreatment Group | Saline Pretreatment Group
Number analyzed (Participants) | 49 | 47
Participants, number | 46 | 30

3. Secondary Outcome: Coughing
Description: Data include patients who coughed irrespective of the degree of coughing.
Time Frame: Intraoperative period
Population: Per protocol
Measure: Number; unit: Participants, number
Arm/Group | Fentanyl Pretreatment Group | Saline Pretreatment Group
Number analyzed (Participants) | 49 | 47
Participants, number | 1 | 6

ADVERSE EVENTS:
Time Frame: Patients were followed for up to 24 hours
Arm/Group | FENTANYL | SALINE
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/47
Other Adverse Events (participants affected / at risk) | 0/49 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No